CLINICAL TRIAL: NCT06433518
Title: What Should Be The Optimal Ovulation Triggering Size in Poseidon Group 4 Patients Undergoing Ovarian Stimulation?
Brief Title: BEst Size for Ovulation Triggering in Poseidon 4 Patients (BEST 4 Study)
Acronym: BEST
Status: Not yet recruiting | Type: Observational
Sponsor: Centrum Clinic IVF Center (Other)
Responsible Party: Principal Investigator, Emre Göksan Pabuçcu, Professor, Centrum Clinic IVF Center
Other Study IDs: 2024-3-1
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Fertilization; Fertilization in Vitro
Keywords: oocyte; IVF; poor responder; ovarian stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women defined as poor responders according to POSEIDON criteria group 4 undergoing IVF: This group of women, who have low serum AMH levels and low antral follicle count obviusly reveal unfavorable ovarian stimulation and reproductive outcomes in daily practice. Since the most important outcome measure is the live birth rate in assisted reproduction, rates have been reportedly very low for this cohort. Depending from the reports, live birth rates particularly cumulative rates directly correlated with collected numbers of oocytes. Therefore, studies should focus on this entity.
  Interventions: Drug: recombinant hCG

INTERVENTIONS:
Drug: recombinant hCG — Experimental Group: Final oocyte triggering will be performed when the follicle or follicles measure between 13-16 mm.
  Control Group: Final oocyte triggering will be performed when the follicle or follicles measure greater than 17 mm.
  All triggers will be administered uniformly with 6500 units of recombinant hCG and 0,2 mg triptorelin injections.
  The primary outcome of the study will be the number of mature oocytes. Secondary outcomes will include fertilization rates, embryo counts, and implantation rates.
  Primary and secondary outcomes will be compared between the two groups.

SUMMARY:
This observational clinical study aims to determine the optimal timing of ovulation triggering in women aged 35 and above with poor ovarian reserve.

For this purpose, cases undergoing ovarian stimulation for assisted reproductive treatment and planned final oocyte triggering will be evaluated in two separate groups:

1. **Experimental Group**: Final oocyte triggering will be performed when the follicle or follicles measure between 13-16 mm.
2. **Control Group**: Final oocyte triggering will be performed when the follicle or follicles measure greater than 17 mm.

All triggers will be administered uniformly with 6500 units of recombinant hCG and 0,2 mg triptorelin injections.

The primary outcome of the study will be the number of mature oocytes. Secondary outcomes will include fertilization rates, embryo counts, and implantation rates.

Primary and secondary outcomes will be compared between the two groups.

DETAILED DESCRIPTION:
The timing of final oocyte maturation in assisted reproductive techniques is critically important. If serum steroid hormone levels are appropriate during the late follicular phase, ovulation triggering can be performed using various agents. There are numerous comparative studies in the literature on this topic.

However, a key issue is determining the most optimal timing for this trigger. In standard practice, the final triggering is performed when the follicle size reaches 17 mm or more.

The purpose of this is to obtain mature eggs from these follicles during the oocyte aspiration process.

However, in some special cases, to maximize the desired yield, this size threshold may be adjusted.

A prime example of this is in older patients with poor ovarian reserve, as the expected egg yield may not be achieved with standard practices.

During the oocyte collection process, fewer mature oocytes (M2) may be retrieved, or no oocytes may be retrieved at all, despite proper ovarian stimulation. Therefore, the optimal follicle size for these cases has not been definitively established in the literature. Thus, there is a need to determine other follicular thresholds specifically for older women with poor ovarian reserves to enhance egg and mature egg yields.

For this purpose, cases undergoing ovarian stimulation for assisted reproductive treatment and planned final oocyte triggering will be evaluated in two separate groups:

1. **Experimental Group**: Final oocyte triggering will be performed when the follicle or follicles measure between 13-16 mm.
2. **Control Group**: Final oocyte triggering will be performed when the follicle or follicles measure greater than 17 mm.

All triggers will be administered uniformly with 6500 units of recombinant hCG and 0,2 mg triptorelin injections.

The primary outcome of the study will be the number of mature oocytes. Secondary outcomes will include fertilization rates, embryo counts, and implantation rates.

Primary and secondary outcomes will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Women age >35 years Women with low serum AMH (<1,2 ng/ml), low AFC (<5) Undergoing assisted reproduction with Short antagonist protocol Max daily gonadotropin dose of 300 IU

Exclusion Criteria:

* women with uterine and/or endometrial abnormality, women with endometrioma(s), short or long GnRH-agonist ovarian stimulation protocols, severe male infertiliy, genetic conditions, with normal ovarian reserve markers, <35 years old, women with prior ovarian surgeries, PGT-a cycles

Ages: 35 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with diminished ovarian reserve undergoing assisted reproduction.
Study Population: A group of women defined as Poseidon Group 4, who will apply to the infertility clinic to be scheduled for ovarian stimulation and assisted conception treatments during the study period.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Mean Mature Oocytes between two triggering strategies | From enrollment to the end of treatment at 6-8 months.
  Mean numbers of oocytes, mature oocytes, fertilization rates, embryos and pregnancy rates will be compared between two different triggering sizes.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Pabuccu, Prof., Study Director — Ufuk University

IPD SHARING:
Plan to Share IPD: No